CLINICAL TRIAL: NCT06652776
Title: The Italian COPD Registry. the DescribinG BUrden of COPD and Occurrence of MortaLity in a Cohort of Italian Patients
Brief Title: The Italian Registry of Patients with Chronic Obstructive Pulmonary Disease
Acronym: ICoRe
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: University of Genova (Other); University of Pavia (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); University Magna Graecia (Other); University of Rome Tor Vergata (Other); Università degli Studi di Sassari (Other); University of Palermo (Other); University of Turin, Italy (Other); University Hospital Verona, Italy (Unknown); University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor, University of Milan
Other Study IDs: 20-27Sept2023
Record Dates: First submitted 2024-09-03; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: COPD; COPD Exacerbation Acute; Comorbid Chronic Lung Disease on Heart Failure; Mortality; Cardiovascular Diseases; Cardiovascular Events; COPD Prevalance
Keywords: COPD; AECOPD; Mortality in AECOPD; COPD mortality risk factors; COPD prevalence; lung function; emphysema; chronic bronchitis; COPD hospitalization; heart failure; cardiovascular mortality; Bronchodilators; COPD therapy; triple therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Emphysema; Bronchitis, Chronic; Heart Failure | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD patients: All patients with a functionally confirmed diagnosis of COPD
  Interventions: Other: Pharmacological treatment

INTERVENTIONS:
Other: Pharmacological treatment — Pharmacological and non pharmacological treatments will be assessed and monitored during the retrospective and prospective phase, and will include:
  * bronchodilators, inhaled steroids and their combinations
  * mucolytics
  * biologic therapies for COPD
  * roflumilast
  * pulmonary rehabilitation
Other: Pharmacological treatment — All pharmacological and non pharmacological treatments for COPD will be assessed and monitored during the retrospective and prospective phase of the study, and will include:
  * inhaled bronchodilators (long term beta-2 agonists and cholinergic antagonists), inhaled corticosteroids and their combinations
  * mucolytics
  * biologics for COPD (monoclonal antibodies)
  * roflumilast
  * chronic oral azythromicin
  * pulmonary rehabilitation
  * oxygen therapy
  * non invasive/invasive ventilation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a treatable but debilitating medical condition associated with persistent symptoms and chronic airflow obstruction. Despite the availability of multiple therapeutic options, COPD is the third leading cause of death worldwide and has a substantial socioeconomic impact.

The present real life study is aimed at describing the clinical and functional characteristics, treatment patterns, impact of exacerbations and comorbidities and their association with mortality in a large cohort of Italian patients with COPD.

DETAILED DESCRIPTION:
The temporal relationship of observation period to time of participant enrollment will be both retrospective and prospective.

A digital dataset will be shared with the participating centers. The following variables, if available, will be collected.

Demographic and clinical variables:

* Age, sex, height, weight, BMI, waist circumference.
* Pneumonia episodes in the last 12 months and number of hospitalizations for pneumonia.
* Number of pulmonary rehabilitation cycles performed
* Vaccination status (Flu, SARS-CoV-2, pneumococcus, human respiratory syncytial virus, herpes zoster)

COPD characteristics:

* Date of COPD diagnosis.
* COPD exacerbations in the year before the index date (mild, moderate, severe exacerbations), hospitalizations and/or access to ICU.
* Type, dosages and duration of antibiotic and systemic corticosteroid treatments during exacerbations.
* Respiratory symptoms evaluated with mMRC and CAT
* Frequency and purulence of sputum, cough frequency
* Inhaled bronchodilator/corticosteroid therapy and type of device used, any treatment changes at index date or during follow up.
* Mucolytic agents (active molecules and dosage)
* Chronic use of azithromycin
* Therapy with roflumilast.
* Biological therapies (type of active molecules, duration, switch).
* Long-term oxygen therapy (FiO2, average flow), presence of tracheostomy and any invasive or non-invasive ventilatory support

Comorbidities:

* Concomitant respiratory diseases, history of exposure to risk factors, smoking history (active, former and non-smoker).
* Cardiovascular comorbidities and complications in the last 12 months before index date and during follow up
* Cardioactive pharmacological therapies
* Charlson score
* Other comorbidities

Biological and functional variables:

* Blood tests (RBC, Hb, hematocrit, MCV, PLT, WBC differential, CRP, glycemia, creatinine, uremia, NT-proBNP, cholesterol).
* Cardiopulmonary exercise test. The variables collected will include: VO2max, WR max, HRmax, VE max, VEmax, VE/VO2 ratio, PET CO2, O2 pulse, anaerobic threshold, A-a gradient. All values will be collected as absolute and as percentage of predicted values.
* Nocturnal oximetry: FiO2, T-90, mean SpO2, ODI.
* Polysomnography: type of support (e.g. CPAP or NIMV), FiO2, apnea-hypopnea index (AHI; obstructive, central, and mixed type), AI, oxygen desaturation index (ODI), T-90, Cheyne-Stokes respiration, snoring and body position during the exam.
* 6 minutes walking test: FiO2, distance walked in meters and predicted value, SpO2 at the beginning and end of the test, desaturation, if SpO2<90, modified Borg dyspnea score at the beginning and end of the test.
* Gas exchange: SpO2, FiO2, Blood Gas Analysis (pH, PaO2, PaCO2, HCO3-, A-a gradient, FiO2, PaO2/FiO2)
* Lung function test pre- and post-bronchodilator: FVC, FEV1, FEV1/FVC, FEF 25-75, VC, IC, FEV1/VC. All values will be collected as absolute values, ratio and percentage of predicted values.
* Body plethysmography pre- and post-bronchodilator: TGV, RV, TLC, RV/TLC, IC/TLC, sRAW. All values will be collected as absolute values, ratio and percentage of predicted values
* Diffusion capacity of the lung for carbon monoxide: DLCO, KCO, VA, TLC/VA
* Fractional exhaled nitric oxide
* Chest imaging: radiography or CT scan, presence of emphysema (panlobular or centrolobular), bronchiectasis or interstitial lung disease.
* Ecocardiography: ejection fraction, pathological signs, PAPs, left ventricular hypertrophy and left atrial, right ventricular or left ventricular enlargement.
* Coronary angiography: if pathological for stenosis and number of involved vessels, PTCA or CABG.

All these items will be also valued during the follow up period, with an emphasis on COPD exacerbations and date and cause of death.

ELIGIBILITY:
Inclusion Criteria:

• established diagnosis of COPD (defined as age ≥ 40 years old, smoking history ≤ 20 pack years, postbronchodilator forced expiratory volume in one second to slow vital capacity ratio (FEV1/VC) ≤ the lower limit of normal (LLN) criteria.

Exclusion Criteria:

* Presence of current clinically significant asthma
* Diagnosis or clinically significant alternative respiratory diseases (such as interstitial lung disease or bronchiectasis)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with functionally confirmed COPD and a track medical record in the 12 months before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | From index date (registry inclusion) until the date of death from any cause, assessed up to 120 months
  Annual all-cause mortality rate
Burden of moderate and severe COPD acute exacerbations | From index date (registry inclusion) until the date of first event of moderate or severe exacerbation, and any following event of moderate or severe exacerbation, or patient's death, whichever comes first, assessed up to 120 months
  Incidence and annual rate of moderate and/or severe exacerbations

SECONDARY OUTCOMES:
Cardiovascular mortality | From index date (registry inclusion) until the date of death provoked by a cardiovascular event, assessed up to 120 months
  Annual death rate for cardiovascular events
Cardiovascular comorbidities | At index date (registry inclusion) comorbidities will be registered and updated at every new visit until patient's death
  prevalence of cardiovascular comorbidities and their relationship with lung function, respiratory symptoms, moderate and severe exacerbations, mortality
Cardiovascular events | From index date (registry inclusion) until the date of any cardiovascular event or cardiovascular death, whichever comes first, assessed up to 120 months
  Incidence and prevalence of cardiovascular events (overall and severe) and their relationship with COPD acute exacerbations
Lung function decline | From index date (registry inclusion) until the date of the first lung function test, and any following available lung function assessment, or the date of patient's death, whichever comes first, assessed up to 120 months
  trend in lung function indexes (spirometric, plethysmographic, DLCO) over time
Eosinophil count | From index date (registry inclusion) until the date of first available eosinophil count, and any following point in time with available eosinophil count updates, or patients' death, whichever comes first, assessed up to 120 months
  Describe eosinophil count in absolute and % of leukocyte formula in the study population, its trend over time and its relationship with lung function, lung function decline, COPD exacerbations, cardiovascular events and mortality
Evaluation of the pharmacological treatment at baseline and treatment switches | From index date (registry inclusion) until the date of first available inhaled treatment switch, and every point in time the patient changes inhaled treatment, or the patient's death from any cause, whichever comes first, assessed up to 120 months
  Prevalence of type of inhaled therapy over time from index date until end of study

OTHER OUTCOMES:
Exacerbation etiology | From index date (registry inclusion) until the date of the first available acute exacerbation of any severity, and any following event of modand any following exacerbation event date, or patient 's death, whichever comes first, assessed up to 120 months
  Describe the frequency and type of viral or bacterial isolates during acute exacerbations, and their relationship with lung function, comorbidities and exacerbation severity
Corticosteroid treatment during COPD exacerbation | From index date (registry inclusion) until the date of first exacerbation of any severity, and any following event of moderate or severe exacerbation, or patient's death, whichever comes first, assessed up to 120 months.
  Describe the frequency and dosage of systemic and oral corticosteroids, treatment duration and their relationship with COPD severity, comorbidities, exacerbation severity and exacerbation etiology
Antibiotic treatments during acute COPD exacerbations | From index date (registry inclusion) until the date of first exacerbation of any severity, and any following event of moderate or severe exacerbation, or patient's death, whichever comes first, assessed up to 120 months.
  Describe the frequency and type of antibiotic treatments, treatment duration and their relationship with COPD severity, comorbidities, exacerbation severity and exacerbation etiology
Gas exchange | From index date (registry inclusion) until the date of first outpatient visit with available data on gas exchange, and any following event (visit) with gas exchange information, or patient's death, whichever comes first, assessed up to 120 months.
  Describe the prevalence of type I and II respiratory failure, trend over time in PaO2 and PaCo2 and their relationship with acute COPD exacerbations, cardiovascular comorbidities, cardiovascular events and mortality
Pneumonia events | From index date (registry inclusion) until the date of first pneumonia event of any severity, and any following event of pneumonia, or patient's death, whichever comes first, assessed up to 120 months.
  incidence and annual pneumonia rate overall and divided by type of patient treatment
Cardiac function | From index date (registry inclusion) until the date of first available cardiac ultrasound, and the date of any following cardiac ultrasound assessment, or patient's death, whichever comes first, assessed up to 120 months.
  Describe cardiac function in terms of heart ultrasound parameters at index date and its relationship with future events such as COPD exacerbations, cardiovascular events and mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Luigi Sacco University Hospital, Division of Department of Biomedical and Clinical Sciences, University of Milan, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santus P, Di Marco F, Braido F, Contoli M, Corsico AG, Micheletto C, Pelaia G, Radovanovic D, Rogliani P, Saderi L, Scichilone N, Tanzi S, Vella M, Boarino S, Sotgiu G, Solidoro P. Exacerbation Burden in COPD and Occurrence of Mortality in a Cohort of Italian Patients: Results of the Gulp Study. Int J Chron Obstruct Pulmon Dis. 2024 Mar 1;19:607-618. doi: 10.2147/COPD.S446636. eCollection 2024. PMID 38444551
- [Background] Radovanovic D, Contoli M, Marco FD, Sotgiu G, Pelaia G, Braido F, Corsico AG, Micheletto C, Rogliani P, Scichilone N, Saderi L, Santus P, Solidoro P. Clinical and Functional Characteristics of COPD Patients Across GOLD Classifications: Results of a Multicenter Observational Study. COPD. 2019 Aug;16(3-4):215-226. doi: 10.1080/15412555.2019.1659760. Epub 2019 Sep 9. PMID 31500459